CLINICAL TRIAL: NCT02705716
Title: Short Term Clinical Study Investigating the Efficacy of an Occluding Dentifrice in Providing Relief From Dentinal Hypersensitivity
Brief Title: Study Investigating Efficacy of an Occluding Dentifrice for Dentine Hypersensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 205212
Record Dates: First submitted 2016-03-07; First posted 2016-03-10 (Estimated); Results first posted 2017-04-25 (Actual); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Dentin Sensitivity
MeSH Terms: conditions — Dentin Sensitivity | interventions — fluorophosphate

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test Dentifrice (Experimental): Participants will be instructed to dose a dry toothbrush with a full strip of toothpaste containing 0.454% weight by weight (w/w) stannous fluoride (1100 parts per million [ppm] fluoride). Participants will then brush each of the two selected sensitive test teeth first, followed by the whole mouth thoroughly for at least 1 minute.
  Interventions: Other: 0.454% w/w stannous fluoride (1100ppm fluoride)
- Control Dentifrice (Placebo Comparator): Participants will be instructed to apply a full brush head of toothpaste containing 0.76% sodium monofluorophosphate (1000ppm fluoride) to a dry toothbrush. Participants will then brush the whole mouth thoroughly for at least 1 minute.
  Interventions: Other: 0.76% sodium monofluorophosphate (1000ppm fluoride)

INTERVENTIONS:
Other: 0.454% w/w stannous fluoride (1100ppm fluoride) — Dentifrice containing 0.454% w/w stannous fluoride (1100ppm fluoride)
  Arms: Test Dentifrice
Other: 0.76% sodium monofluorophosphate (1000ppm fluoride) — Dentifrice containing 0.76% sodium monofluorophosphate (1000ppm fluoride)
  Arms: Control Dentifrice

SUMMARY:
This study will investigate the efficacy of an experimental dentifrice containing 0.454% weight/weight (w/w) stannous fluoride in relieving dentine hypersensitivity (DH) after twice daily brushing, over a 2 week treatment period compared with a standard fluoride dentifrice.

ELIGIBILITY:
Inclusion Criteria:

* Demonstrates understanding of the study procedures, restrictions and willingness to participate as evidenced by voluntary written informed consent and has received a signed and dated copy of the informed consent form.
* Participant is male or female aged between 18 and 65 years inclusive.
* Good general and mental health with, in the opinion of the investigator or medically qualified designee.
* No clinically significant and relevant abnormalities in medical history or upon oral examination.
* Absence of any condition that would impact on the participant's safety or well being or affect the individual's ability to understand and follow study procedures and requirements.
* Self-reported history of dentinal hypersensitivity (DH) lasting more than(>) six months but not > 10 years.
* Good general oral health, with a minimum of 20 natural teeth.
* Minimum of 2 accessible non-adjacent teeth (incisors, canines, pre-molars), preferably in different quadrants at screening and minimum of two, non-adjacent accessible teeth (incisors, canines, pre-molars) at baseline.

Exclusion Criteria:

* Women who are pregnant or breast-feeding .
* Daily doses of medication/treatments which, in the opinion of the Investigator, could interfere with the perception of pain. Examples of such medications include analgesics, anticonvulsants, antihistamines that cause marked or moderate sedation, sedatives, tranquilisers, anti-depressants, mood-altering and anti-inflammatory drugs.
* Currently taking antibiotics or has taken antibiotics within two weeks of Baseline.
* Daily dose of a medication which, in the opinion of the investigator, is causing xerostomia.
* Presence of kidney disease, hyperoxaluria, or any other condition that may be exacerbated by oxalic acid or oxalate salts.
* Presence of chronic debilitating disease which, in the opinion of the investigator, could affect study outcomes.
* Any condition which, in the opinion of the investigator, causes xerostomia.
* Known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients.
* Participation in another clinical study (including cosmetic studies) or receipt of an investigational drug within 30 days of the screening visit.
* Previous participation in this study.
* Recent history (within the last year) of alcohol or other substance abuse.
* Dental prophylaxis within four weeks of Screening, tongue or lip piercing or presence of dental implants.
* Desensitizing treatment within eight weeks of Screening (professional sensitivity treatments and non-toothpaste sensitivity treatments).
* Gross periodontal disease, treatment of periodontal disease (including surgery) within 12 months of Screening, scaling or root planning within 3 months of Screening.
* Teeth bleaching within eight weeks of Screening.
* Tooth with evidence of current or recent caries, or reported treatment of decay within 12 months of Screening.
* Tooth with exposed dentine but with deep, defective or facial restorations, teeth used as abutments for fixed or removable partial dentures, teeth with full crowns or veneers, orthodontic bands or cracked enamel. Sensitive teeth with contributing aetiologies other than erosion, abrasion or recession of exposed dentine.
* Sensitive tooth not expected to respond to treatment with an over-the-counter toothpaste in the opinion of the Investigator.
* Use of an oral care product indicated for the relief of dentine hypersensitivity within eight weeks of screening.
* Individuals who require antibiotic prophylaxis for dental procedures.
* Any participant who, in the judgment of the investigator, should not participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 409 (Actual)
Dates: Start 2016-03-01; Primary Completion 2016-05-20 (Actual); Study Completion 2016-05-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- United Kingdom (3):
  - GSK Investigational Site, Ellesmere Port, Cheshire
  - GSK Investigational Site, Manchester
  - GSK Investigational Site, Metropolitan Borough of Wirral

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at one center (2 sites) in United Kingdom.
Pre-assignment Details: A total of 409 participants were screened, out of which 142 participants were randomized. 267 participants were not randomized because 183 participants did not met the study criteria, 1 had adverse event, 2 were lost to follow up, 7 had protocol violation, 2 withdrew consent and 72 were not randomized for other reasons (not specified).
Groups:
- Test Dentifrice: Participants were instructed to dose a dry toothbrush with a full strip of test dentifrice containing 0.454% weight by weight (w/w) stannous fluoride (1100 parts per million [ppm] fluoride). Participants then brushed each of the two selected sensitive test teeth first, followed by the whole mouth thoroughly for at least 1 minute. Participants were permitted to rinse with tap water after brushing.
- Control Dentifrice: Participants were instructed to apply a full brush head of control dentifrice containing 0.76% sodium monofluorophosphate (1000ppm fluoride) to a dry toothbrush. Participants then brushed the whole mouth thoroughly for at least 1 minute. Participants were permitted to rinse with tap water after brushing.
Period: Overall Study
Arm/Group | Test Dentifrice | Control Dentifrice
Started | 72 | 70
Completed | 68 | 68
Not Completed | 4 | 2
Not completed — Adverse Event | 0 | 1
Not completed — Protocol Violation | 3 | 0
Not completed — Withdrawal of Consent | 1 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all the participants who were randomized, received at least one dose of the study treatment and provided at least one post-baseline assessment of efficacy.
Groups:
- Test Dentifrice: Participants were instructed to dose a dry toothbrush with a full strip of test dentifrice containing 0.454% w/w stannous fluoride (1100 ppm fluoride). Participants then brushed each of the two selected sensitive test teeth first, followed by the whole mouth thoroughly for at least 1 minute. Participants were permitted to rinse with tap water after brushing.
- Control Dentifrice: Participants were instructed to apply a full brush head of control dentifrice containing 0.76% w/w sodium monofluorophosphate (1000ppm fluoride) to a dry toothbrush. Participants then brushed the whole mouth thoroughly for at least 1 minute. Participants were permitted to rinse with tap water after brushing.
- Total: Total of all reporting groups
Arm/Group | Test Dentifrice | Control Dentifrice | Total
Number analyzed (Participants) | 70 | 69 | 139
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.9 (10.72) | 39.9 (9.53) | 39.9 (10.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 57 | 110
  Male | 17 | 12 | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 68 | 69 | 137
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 7 | 14
  White | 57 | 59 | 116
  More than one race | 3 | 0 | 3
  Unknown or Not Reported | 0 | 0 | 0
Schiff Sensitivity Score at Baseline [Mean (Standard Deviation); unit: score on a scale] — Assessed by examiner as participant's response to an evaporative (air) stimulus after stimulation of each individual tooth, scored using Schiff sensitivity scale range of 0-3; 0=Participant does not respond to air stimulation; 1=Participant responds to air stimulus but does not request discontinuation of stimulus; 2=Participant responds to air stimulus & requests discontinuation or moves from stimulus; 3=Participant responds to stimulus, considers stimulus to be painful, & requests discontinuation of stimulus. A reduction in Schiff Sensitivity score indicates improvement in sensitivity. Population: This baseline measurement was performed on intent to treat (ITT) population, defined as all participants who were randomized, received study treatment at least once & provided at least one post-baseline (post treatment) assessment of efficacy.
  score on a scale | 2.80 (0.323) | 2.83 (0.307) | 2.81 (0.314)
Tactile Threshold at Baseline [Mean (Standard Deviation); unit: gram (g)] — Tactile threshold was assessed by examiner using a constant pressure probe (Yeaple probe) which allowed application of a known force to the dentin surface from 10 g to an upper threshold of 80g in increments of 10 g. Tactile threshold is the maximum pressure applied at which participant do not report any pain or discomfort. Tactile threshold for each tooth was determined by asking participant whether sensation caused discomfort. The pressure setting at which participant gave two consecutive 'yes' responses was recorded as tactile threshold. Higher tactile threshold, less sensitive tooth. Population: This baseline measurement was performed on ITT population, defined as all participants who were randomized, received study treatment at least once & provided at least one post-baseline (post treatment) assessment of efficacy.
  gram (g) | 11.50 (2.739) | 12.03 (3.010) | 11.76 (2.878)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Schiff Sensitivity Score on Day 14
Description: Schiff sensitivity score was assessed by examiner as participant's response to an evaporative (air) stimulus after the stimulation of each individual tooth. Response of participant was scored using Schiff sensitivity scale range of 0-3; 0=Participant does not respond to air stimulation; 1=Participant responds to air stimulus but does not request discontinuation of stimulus; 2=Participant responds to air stimulus and requests discontinuation or moves from stimulus; 3= Participant responds to stimulus, considers stimulus to be painful, and requests discontinuation of the stimulus. A reduction in Schiff Sensitivity score indicates improvement in sensitivity.
Time Frame: Baseline, Day 14
Population: Analysis for this outcome was conducted on ITT population, defined as all participants who were randomized, received study treatment at least once & provided at least one post-baseline (post treatment) assessment of efficacy. Number of participants analyzed is number of participants from ITT population evaluated on Day 14.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Test Dentifrice | Control Dentifrice
Number analyzed (Participants) | 68 | 68
score on a scale | -1.01 (1.093) | -0.88 (1.110)
Statistical Analysis 1: Comparison: Test Dentifrice vs Control Dentifrice; Test type: Other; p = 0.5191, ANCOVA; From ANCOVA Model, Response: change from baseline in Schiff sensitivity score Factors: treatment & site Covariates: baseline Schiff sensitivity score; Least Square (LS) Mean Difference = -0.12, 95% CI 2-sided [-0.497 to 0.252] — Difference is first named dentifrice minus second named dentifrice such that a negative difference favors first named dentifrice

2. Secondary Outcome: Change From Baseline in Schiff Sensitivity Score on Day 7
Description: as for outcome 1
Time Frame: Baseline, Day 7
Population: Analysis for this outcome was conducted on ITT population, defined as all participants who were randomized, received study treatment at least once & provided at least one post-baseline (post treatment) assessment of efficacy. Number of participants analyzed is number of participants from ITT population evaluated on Day 7.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Test Dentifrice | Control Dentifrice
Number analyzed (Participants) | 70 | 69
score on a scale | -0.49 (0.807) | -0.54 (0.785)

3. Secondary Outcome: Change From Baseline in Tactile Threshold on Day 7 and 14
Description: Tactile threshold was assessed by examiner using a constant pressure probe (Yeaple probe) which allowed application of a known force to the dentin surface from 10 g to an upper threshold of 80g in increments of 10 g. The tactile threshold is the maximum pressure applied at which participant do not report any pain or discomfort. The tactile threshold for each tooth was determined by asking the participant whether the sensation caused discomfort. The pressure setting at which the participant gave two consecutive 'yes' responses was recorded as the tactile threshold. The higher the tactile threshold, the less sensitive the tooth.
Time Frame: Baseline, Day 7 and Day 14
Population: Analysis for this outcome was conducted on ITT population, defined as all participants who were randomized, received the study treatment at least once and provided at least one post-baseline (post treatment) assessment of efficacy. n=number of participants evaluated at specific time points for each treatment arms respectively.
Measure: Mean (Standard Deviation); unit: g
Arm/Group | Test Dentifrice | Control Dentifrice
Number analyzed (Participants) | 70 | 69
g
  Change from baseline on Day 7(n=70,69) | 11.21 (19.531) | 10.29 (17.634)
  Change from baseline on Day 14(n=68,68) | 18.24 (24.522) | 18.90 (23.081)

ADVERSE EVENTS:
Arm/Group | Test Dentifrice | Control Dentifrice
All-Cause Mortality (participants affected / at risk) | 0/72 | 0/70
Serious Adverse Events (participants affected / at risk) | 0/72 | 0/70
Other Adverse Events (participants affected / at risk) | 15/72 | 10/70
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Test Dentifrice (N=72) | Control Dentifrice (N=70)
Food Poisoning (Gastrointestinal disorders) | 1 | 0
Gingival Discomfort (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Noninfective Gingivitis (Gastrointestinal disorders) | 1 | 0
Oral Mucosal Exfoliation (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 1
Ligament Sprain (Injury, poisoning and procedural complications) | 2 | 0
Traumatic Ulcer (Injury, poisoning and procedural complications) | 2 | 1
Procedural Pain (Injury, poisoning and procedural complications) | 1 | 0
Tooth Fracture (Injury, poisoning and procedural complications) | 1 | 0
Conjunctivitis (Infections and infestations) | 1 | 2
Gastroenteritis (Infections and infestations) | 1 | 0
Oral Herpes (Infections and infestations) | 1 | 1
Rhinitis (Infections and infestations) | 1 | 1
Sepsis (Infections and infestations) | 1 | 0
Root Canal Infection (Infections and infestations) | 0 | 1
Device Failure (Product Issues) | 1 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rash Generalised (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.